CLINICAL TRIAL: NCT05037071
Title: The Impact of Upper Body Compression Wear on Muscle Tissue Oxygen Saturation During Video Game Play in Competitive Gamers.
Brief Title: Arm Compression on Muscle Oxygen Saturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Joanne DiFrancisco-Donoghue, Associate Professor, New York Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: BHS-1674
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Muscle; Fatigue, Heart
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Upper body compression (Experimental): An arm compression sleeve with a graduated compression between 18-25 mmHg will be worn on the dominant gaming arm while performing intense gridlock training using an AIM trainer lab. Muscle oxygen saturation of the extensor radialis muscle will be measured using near infrared spectroscopy.
  Interventions: Device: Upper body graduated compression sleeve
- No compression (No Intervention): Muscle oxygen saturation of the extensor radialis muscle will be measured using near infrared spectroscopy on the dominant gaming arm while performing intense gridlock training using an AIM trainer lab. .

INTERVENTIONS:
Device: Upper body graduated compression sleeve — An over the counter light compression sleeve will be worn during game training
  Arms: Upper body compression

SUMMARY:
This study is designed to observe muscle oxygen saturation during intense video game using gridlock training with and without upper arm compression sleeves.

DETAILED DESCRIPTION:
A competitive esport player can perform up to 500-600 mouse and keyboard actions per minute (APM) on a typical training day. A routine training day for a competitive esport player can range from 5- 10 hours of play with no break. In comparison, office workers perform an average of 130-180 keyboard and mouse inputs over the course of an 8 hour work day. These APM's require sustained wrist extension in conjunction with repetitive forearm muscle contractions in multiple planes, as well as shoulder stability and postural stability.

Maneuvering a mouse and keyboard requires repeated contractions of the extensor carpi ulnaris and extensor digitorum. With these fine motor demands, it is common for players to suffer from acute and chronic overuse wrist and arm injuries.

Muscle tissue oxygenation (Sm02) saturation is important to all athletic populations including endurance athletes and power athletes. It's a marker of how efficient that muscle is performing. A decrease in Sm02 indicates less ATP to that muscle and fatigue. Muscle deoxygenation and reoxygenation has been studied in multiple athletic populations. In competitive rock climbers, a lesser rate of deoxygenation of the finger and wrist extensor muscles was related to a higher level of climbing ability.

The use of compression wear has expanded from clinical use into the sports market. The recommendations to wear compression gear in athletes is based on improvement in venous blood flow which improves exchange of fresh blood and blood waste. The research on its use on improving running performance has been mixed. Anecdotally, in 2001 Allen Iverson of the National Basketball Association (NBA) wore a compression arm sleeve to prevent swelling and provide relief of bursitis in his elbow. Lebron James of the NBA and London marathon runner Paul Radcliffe both swear by compression gear. In the 2016 Olympics, it was estimated that 90% of athletes used some form of compression performance gear. The compression wear sports industry market is a billion-dollar industry projected to be worth 3.96 billion dollars by 2022.

Athletes in various sports wear compression garments with the assumption that it will improve performance and facilitate muscle recovery. Most modern compression gear marketed toward athletes use 'graduated compression'. This means that the highest amount of pressure is on the most distal parts of your body (e.g ankles if you are using lower body compression) and the pressure gradually reduces as it moves up toward your body. Compression wear varies in pressure range. The measurement is measured in mmHg and light compression can range from 18-21 mmHg, moderate 23-32 mmHg, strong 34-46 mmHg and > 49 mmHg very strong. (6) Most over the counter athletic compression garments range from 18-21 mmHg.

With esports literature in its infant stages, oxidative capacity of the finger and wrist extensors during prolonged gaming have never been explored. The aim of this study is to compare changes in tissue oxygenation of the wrist extensor muscles with and without graduated arm compression during competitive game play.

ELIGIBILITY:
Inclusion Criteria:

* A ranked esport player with over 500 hours in your game
* Non-smoker
* No history of heart disease
* No history of pulmonary disease
* No history of metabolic disease including diabetes

Exclusion Criteria:

-taking any prescribed or over the counter medications that would influence metabolic outcomes or blood viscosity.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Muscle tissue oxygen saturation | 30 minutes
  A MOXY muscle oxygen sensor will be used on the extensor carpi radialis longus muscle to measure how much muscle desaturation occurs while playing video games that require a mouse.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donoghue, Principal Investigator — Director of Clinical Research
Locations (1):
- New York Institute of Technology College of Osteopathic Medicine, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DiFrancisco-Donoghue J, Rothstein A, Jung MK, Zwibel H, Werner WG. Upper body compression wear improves muscle oxygenation following intense video game training: a randomized cross-over study among competitive gamers. BMC Sports Sci Med Rehabil. 2023 Sep 11;15(1):108. doi: 10.1186/s13102-023-00720-5. PMID 37697389